CLINICAL TRIAL: NCT06691048
Title: Descriptive Study of Adult Patients Diagnosed Later with a Neurodevelopmental Disorder and Their Management
Brief Title: Neurodevelopmental Disorder Diagnosis During Adulthood
Acronym: NeuroDevAD
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_5397
Record Dates: First submitted 2024-05-17; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Neurodevelopmental Disorders
Keywords: Neurodevelopmental Disorders; Late diagnosis; Adult
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults with late diagnosis neurodevelopmental disorder: Adults with late access to diagnosis of neurodevelopmental disorder
  Interventions: Other: Description of an adult population diagnosed late with a neurodevelopmental disorder

INTERVENTIONS:
Other: Description of an adult population diagnosed late with a neurodevelopmental disorder — Clinical description during diagnostic interview

SUMMARY:
The prevalence of neurodevelopmental disorders (specific learning disorders: dyslexia, dysorthographia, dysgraphia and dyscalculia; communication disorders; developmental coordination disorders; attention deficit disorder with or without hyperactivity (ADHD); intellectual disability (ID) and autism spectrum disorders) in the general population is very high, representing over 15% of the paediatric population. Among this population, between 40% and 90% remain symptomatic into adulthood. In addition to the part of the population diagnosed in childhood and lost to the transition to adulthood, a significant part of this population remains unidentified and therefore untreated (up to 60%). It is in adulthood that the diagnosis of neurodevelopmental disorders must be identified as being at the origin of at least some of the cognitive dysfunctions observed: failure at school, difficulties in socio-professional integration... Thus, the lifelong care diagnostic pathway needs to be developed both from an organizational point of view and in terms of the scientific knowledge required to best organize a personalized health pathway for this population. The current challenge for this population is to offer a structured care pathway, from diagnosis to care and medico-social integration.

This project will provide comprehensive, homogeneous data for cohorts of patients requiring diagnostic advice and lifelong management of their disorders. Thesecomprehensive data will contribute to scientific publications on patient cohorts. At present, very few centers have complete, homogeneous data on late-diagnosis adults, so our project will have a scientific and academic impact in its own right.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 or over
* Men or women under 55 years of age
* Patients with a neurodevelopmental disorder according to the latest DSM5 criteria diagnosed after age 18
* Patient with sufficient visual and auditory skills, oral and written language in French accessible to clinical and neuropsychological evaluation.

Exclusion Criteria:

* Patients with intellectual disabilities
* Patients with serious addictive and/or psychiatric comorbidities

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 300 subjects with one or more neurodevelopmental disorders of late diagnosis (i.e. diagnosed in adulthood), with access to a diagnostic opinion in the neurological hospital's functional neurology and epileptology department, between January 2022 and the end of 2024.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Characteristics in Late-Diagnosed Adults with Neurodevelopmental Disorders | At the inclusion
  Social Data: Number of participants with specified social characteristics (e.g., employment status, living arrangements, education level).
Clinical Characteristics in Late-Diagnosed Adults with Neurodevelopmental Disorders | At the inclusion
  Environmental Data: Number of participants with specified environmental factors (e.g., access to care, socioeconomic status).
Clinical Characteristics in Late-Diagnosed Adults with Neurodevelopmental Disorders | At the inclusion
  Health Data: Number of participants with specific health characteristics (e.g., comorbid conditions, history of mental health support, medication use).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No